CLINICAL TRIAL: NCT00911612
Title: A Phase IIB Study to Evaluate the Effects of Welchol (Colesevelam Hydrochloride) on Colonic Transit, Intestinal Permeability and Bowel Function in Diarrhea-predominant Irritable Bowel Syndrome (D-IBS)
Brief Title: Does Welchol (Colesevelam Hydrochloride) Improve Colonic Transit in Diarrhea-predominant Irritable Bowel Syndrome (D-IBS)?
Acronym: welchol
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Mayo Clinic (Other)
Collaborators: National Institute of Diabetes and Digestive and Kidney Diseases (NIDDK) (NIH)
Responsible Party: Michael Camilleri, M.D., Mayo Clinic
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 08-007454; R01DK054681 (NIH)
Record Dates: First submitted 2009-05-29; First posted 2009-06-02 (Estimated); Results first posted 2012-03-15 (Estimated); Last update posted 2012-04-04 (Estimated); Status verified 2012-03

CONDITIONS: Irritable Bowel Syndrome; Diarrhea
Keywords: bile acid; malabsorption; permeability; diarrhea; IBS; stool
MeSH Terms: conditions — Irritable Bowel Syndrome; Diarrhea; Malabsorption Syndromes | interventions — Colesevelam Hydrochloride

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Colesevelam (Experimental): Participants received colesevelam 1.875 g twice daily
  Interventions: Drug: Colesevelam
- Placebo (Placebo Comparator): Participants received an inert capsule matching the study drug twice daily, as prepared by the Mayo Clinic research pharmacy
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Colesevelam — Welchol (Colesevelam HCL) 1.875 gram twice daily for 12-14 days
  Other Names: Welchol
  Arms: Colesevelam
Drug: Placebo — Inert capsule matching the study drug, given twice daily
  Arms: Placebo

SUMMARY:
Our hypothesis is that the medication approved for treatment of high blood cholesterol levels, Colesevelam HCl (WELCHOL), decreases colonic transit and permeability in patients with diarrhea due to irritable bowel syndrome.

This effect is thought to result from the effect of the medication on bile acids, which can cause diarrhea.

DETAILED DESCRIPTION:
Background:

Irritable bowel syndrome (IBS) affects about 15% of the U.S. population, about 5% having predominant diarrhea; current treatment is suboptimal as it may not be tolerated, lead to side effects or insufficient benefit. Bile acid malabsorption (BAM) is recognized as a cause of chronic diarrhea and has been investigated as a mechanism for the phenotype of diarrhea predominant IBS (D-IBS). Increased exposure of the colon to bile acids which may result from accelerated small bowel transit or abnormal function of the apical sodium bile acid transporter (ASBT) has been postulated to cause functional diarrhea or symptoms of D-IBS by a number of mechanisms, such as increase colonic secretion, and mucosal permeability. Recent preliminary data suggest that doses of chenodeoxycholate (CDC) that are approved for the dissolution of gall stones are associated with accelerated colonic emptying and looser stool consistency.

Hypothesis:

The bile acid binding agent, Colesevelam HCl, decreases colonic transit and permeability in patients with D-IBS.

Specific Aim:

To investigate the effect of Colesevelam, which binds bile acids in the small intestine and reduces the concentration of bile acids in the colon, on colonic transit, permeability and the bowel function of patients with D-IBS.

Methods:

Twenty-four D-IBS participants will be randomized to placebo or treatment with Welchol (Colesevelam HCL) 1.875 gram b.i.d. for 12-14 days. A baseline colon transit, 24 hour urine for colon permeability, and blood for serum 7 alpha-hydroxy-4-cholesten-3-one (7 alpha-HCO) will be measured and venous blood DNA will be collected and stored. The measurement of serum 7 alpha-hydroxy-4-cholesten-3-one (7 alpha-HCO), which is a measurement of hepatic cholesterol synthesis, is closely related to the fecal loss of bile acids, and is a validated method for screening for BAM. Following treatment for 12 days, transit and permeability studies will be repeated. Bowel function symptoms will be recorded for the duration of the study.

ELIGIBILITY:
Inclusion Criteria:

* Patients with D-IBS
* Aged 18-65 years
* No abdominal surgery (except appendectomy or cholecystectomy as long as patients IBS-diarrhea symptoms preceded the cholecystectomy

Exclusion Criteria:

* Participants with known chronic liver disease or Aspartate aminotransferase (AST) or Alanine transaminase (ALT) > 2.0 X upper limit of normal
* Hypertriglyceridemia and pancreatitis by history
* Diabetes or hypoglycemia
* Significant coagulation disorder
* History of bowel obstruction
* Serum triglycerides >500 mg/dL
* History of vitamin A, D, E, or K deficiencies

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 24 (Actual)
Dates: Start 2009-01; Primary Completion 2009-05 (Actual); Study Completion 2009-05 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Michael L. Camilleri, M.D., Principal Investigator — Mayo Clinic
Locations (1):
- Mayo Clinic, Rochester, Minnesota, United States

REFERENCES:
- [Background] Fernandez-Banares F, Esteve M, Salas A, Alsina M, Farre C, Gonzalez C, Buxeda M, Forne M, Rosinach M, Espinos JC, Maria Viver J. Systematic evaluation of the causes of chronic watery diarrhea with functional characteristics. Am J Gastroenterol. 2007 Nov;102(11):2520-8. doi: 10.1111/j.1572-0241.2007.01438.x. Epub 2006 Aug 4. PMID 17680846
- [Result] Odunsi-Shiyanbade ST, Camilleri M, McKinzie S, Burton D, Carlson P, Busciglio IA, Lamsam J, Singh R, Zinsmeister AR. Effects of chenodeoxycholate and a bile acid sequestrant, colesevelam, on intestinal transit and bowel function. Clin Gastroenterol Hepatol. 2010 Feb;8(2):159-65. doi: 10.1016/j.cgh.2009.10.020. Epub 2009 Oct 30. PMID 19879973

RESULTS

PARTICIPANT FLOW:
Recruitment Details: All participants were recruited from the Mayo Clinic in Rochester, Minnesota from January through May 2009. 31 subjects signed consent, 1 withdrew consent before the start of the study, 2 had concomitant illness and 4 did not qualify based on colon transit eligibility criteria. 24 subjects were randomized and were included in the analysis.
Period: Overall Study
Arm/Group | Colesevelam | Placebo
Started | 12 | 12
Completed | 12 | 12
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Colesevelam | Placebo | Total
Number analyzed (Participants) | 12 | 12 | 24
Age Continuous [Mean (Standard Deviation); unit: years] | 42.1 (4.0) | 43.3 (3.7) | 42.8 (13.0)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 12 | 12 | 24
  Male | 0 | 0 | 0
Region of Enrollment [Number; unit: participants]
  United States | 12 | 12 | 24
Body Mass Index [Mean (Standard Deviation); unit: kg/m^2] | 31.8 (1.5) | 28.9 (1.8) | 30.4 (5.7)
Baseline Colonic Geometric Center at 24 hours [Mean (Standard Deviation); unit: units on a scale] — The scintigraphic method is used to measure colonic transit. An isotope is adsorbed on activated charcoal particles and delivered to the colon in a delayed release capsule. Anterior and posterior gamma images are taken hourly. The geometric center (GC) is the weighted average of counts in the different colonic regions. The scale ranges from 1 to 5; a high GC implies faster colonic transit. A GC of 1 implies all isotope is in the ascending colon, and a GC of 5 implies all isotope is in the stool.
  units on a scale | 3.4 (0.3) | 3.4 (0.3) | 3.4 (0.2)
Fasting Serum 7 alpha-HCO [Mean (Standard Deviation); unit: ng/mL] — The measurement of serum 7 alpha-hydroxy-4-cholesten-3-one (7 alpha-HCO) is a measurement of hepatic cholesterol synthesis, is closely related to the fecal loss of bile acids, and is a validated method for screening for bile acid malabsorption (BAM).
  ng/mL | 31.8 (5.9) | 38.2 (14.7) | 35.0 (36.5)

OUTCOME MEASURES:

1. Primary Outcome: Colonic Transit, Geometric Center at 24 Hours
Description: The scintigraphic method is used to measure colonic transit. An isotope is adsorbed on activated charcoal particles and delivered to the colon in a delayed release capsule. Anterior and posterior gamma images are taken hourly. The geometric center (GC) is the weighted average of counts in the different colonic regions. The scale ranges from 1 to 5; a high GC implies faster colonic transit. A GC of 1 implies all isotope is in the ascending colon, and a GC of 5 implies all isotope is in the stool.
Time Frame: After 12-14 days treatment
Measure: Mean (Standard Error); unit: units on a scale
Arm/Group | Colesevelam | Placebo
Number analyzed (Participants) | 12 | 12
units on a scale | 2.68 (0.32) | 3.30 (0.33)
Statistical Analysis 1: Comparison: Colesevelam vs Placebo; An analysis of covariance was used to compare drug with placebo adjusting for baseline geometric center at 24 hours , BMI, and 7 alpha CHO; Test type: Superiority or Other; p = 0.22, ANCOVA — Not adjusted since only one comparison was made

2. Primary Outcome: Ascending Colon Emptying T1/2
Description: The half time for the ascending colon emptying (T1/2) was measured by the scintigraphic method. An isotope is adsorbed on activated charcoal particles and delivered to the colon in a delayed release capsule that is swallowed by the subject. Anterior and posterior gamma images are taken hourly. From the hourly scans, a time-activity curve is plotted using linear interpolation between time points when content was measured. The time taken to empty 50% of the isotope from the ascending colon is read from this time-activity curve.
Time Frame: After 12-14 days' treatment
Measure: Mean (Standard Error); unit: hours
Arm/Group | Colesevelam | Placebo
Number analyzed (Participants) | 12 | 12
hours | 18.85 (2.88) | 14.9 (3.58)
Statistical Analysis 1: Comparison: Colesevelam vs Placebo; An analysis of covariance was used to compare drug with placebo adjusting for BMI and 7 alpha HCO; Test type: Superiority or Other; p = 0.02, ANCOVA

3. Secondary Outcome: Colonic Permeability as Measured by Cumulative Urinary Excretion of Mannitol 8-24 Hours
Description: Colonic permeability is measured through differential excretion of urine saccharides. The subject ingests a methacrylate-coated capsule that contains saccharides (mannitol 1g and lactulose 5 g powder). The capsule provides a means to protect the sugars from absorption, until the sugars are delivered to the colon by means of a standard delayed release capsule. The value reported is the mean for each arm of the total amount of mannitol excreted over the 8-24 hour time period.
Time Frame: after 12-14 days' treatment
Measure: Mean (Standard Error); unit: mg
Arm/Group | Colesevelam | Placebo
Number analyzed (Participants) | 12 | 12
mg | 64.3 (13.3) | 45.8 (8.8)

4. Secondary Outcome: Colonic Transit, Geometric Center at 48 Hours
Description: as for outcome 1
Time Frame: After 12-14 days' treatment
Measure: Mean (Standard Error); unit: units on a scale
Arm/Group | Colesevelam | Placebo
Number analyzed (Participants) | 12 | 12
units on a scale | 4.65 (0.13) | 4.47 (0.20)

5. Secondary Outcome: Stool Consistency
Description: The subjects rated their stool consistency using the Bristol Stool Scale. The Bristol Stool Scale is a medical aid designed to classify the form of human feces into seven categories or types. Types 1 and 2 indicate constipation with 3 and 4 being the "ideal stools" especially the latter, as they are the easiest to defecate, and 5-7 tending towards diarrhea.
Time Frame: After 12-14 days' treatment
Measure: Mean (Standard Error); unit: units on a scale
Arm/Group | Colesevelam | Placebo
Number analyzed (Participants) | 12 | 12
units on a scale | 3.78 (0.27) | 4.57 (0.35)

ADVERSE EVENTS:
Time Frame: Adverse events were collected from randomization through the 12-14 day treatment period (colesevelam HCL or placebo) and the 2 day testing period.
Arm/Group | Colesevelam | Placebo
Serious Adverse Events (participants affected / at risk) | 0/12 | 0/12
Other Adverse Events (participants affected / at risk) | 12/12 | 9/12
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Colesevelam (N=12) | Placebo (N=12)
Uterine cramps (Reproductive system and breast disorders) | 1 (1) | 2 (2)
Headache (Nervous system disorders) | 5 (5) | 4 (4)
Upper respiratory infection (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 4 (4)
Lower abdominal cramps (Gastrointestinal disorders) | 2 (2) | 0 (0)
Flatulence (Gastrointestinal disorders) | 3 (3) | 1 (1)
Green-colored stools (Gastrointestinal disorders) | 2 (2) | 2 (2)
Nausea (Gastrointestinal disorders) | 2 (2) | 3 (3)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes; Agreement restricts PI disclosure of results: No